CLINICAL TRIAL: NCT04736173
Title: Official Title: A Phase 2 Study to Evaluate Zimberelimab (AB122) Combined With AB154 in Front-Line, PD-L1-High, Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Study Evaluating Effectiveness and Safety of Zimberelimab and Domvanalimab in Lung Cancer
Acronym: ARC-10
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARC-10; 2020-003562-39 (EudraCT Number); PHRR210222-003371 (Other: Philippine Health Research Registry); 2022-503071-28-00 (EU CTIS Number)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer; Nonsquamous Non Small Cell Lung Cancer; Squamous Non Small Cell Lung Cancer; Lung Cancer
Keywords: Domvanalimab; Zimberelimab; Non Small Cell Lung Cancer; Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — zimberelimab; Carboplatin; Paclitaxel; Pemetrexed; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A - Study Part 1 (Platinum-based Chemotherapy) (Active Comparator): Participants will receive carboplatin, pemetrexed, and paclitaxel by intravenous (IV) infusion.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed
- Arm B - Study Part 1 (Zimberelimab Monotherapy) (Experimental): Participants will receive zimberelimab monotherapy by IV infusion.
  Interventions: Drug: Zimberelimab
- Arm C - Study Part 1 (Domvanalimab + Zimberelimab Combination Therapy) (Experimental): Participants will receive zimberelimab in combination with AB154 by IV infusion.
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- Arm D - Study Part 2 (Domvanalimab + Zimberelimab Combination Therapy) (Experimental): Participants will receive domvanalimab in combination with zimberelimab by IV infusion.
  Interventions: Drug: Domvanalimab; Drug: Zimberelimab
- Arm E - Study Part 2 (Pembrolizumab) (Active Comparator): Participants will receive pembrolizumab by IV infusion.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Domvanalimab — Domvanalimab is a humanized monoclonal antibody targeting human TIGIT
  Other Names: AB154
  Arms: Arm C - Study Part 1 (Domvanalimab + Zimberelimab Combination Therapy); Arm D - Study Part 2 (Domvanalimab + Zimberelimab Combination Therapy)
Drug: Zimberelimab — Zimberelimab is a fully human anti-PD-1 monoclonal antibody
  Other Names: AB122
  Arms: Arm B - Study Part 1 (Zimberelimab Monotherapy); Arm C - Study Part 1 (Domvanalimab + Zimberelimab Combination Therapy); Arm D - Study Part 2 (Domvanalimab + Zimberelimab Combination Therapy)
Drug: Carboplatin — Participants receive carboplatin, pemetrexed, and paclitaxel at a target area under the curve.
  Arms: Arm A - Study Part 1 (Platinum-based Chemotherapy)
Drug: Paclitaxel — Participants receive carboplatin, pemetrexed, and paclitaxel at a target area under the curve.
  Arms: Arm A - Study Part 1 (Platinum-based Chemotherapy)
Drug: Pemetrexed — Participants receive carboplatin, pemetrexed, and paclitaxel at a target area under the curve.
  Arms: Arm A - Study Part 1 (Platinum-based Chemotherapy)
Drug: Pembrolizumab — Pembrolizumab is a humanized Immunoglobulin G4 monoclonal antibody targeting the PD-1 receptor
  Arms: Arm E - Study Part 2 (Pembrolizumab)

SUMMARY:
This is a phase 2 study to evaluate zimberelimab (AB122) combined with domvanalimab (AB154) in front-line, PD-L1-high, locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed, treatment naïve, locally advanced or metastatic (stage IIIB IV per AJCC version 8), squamous or non-squamous NSCLC with documented high PD L1 expression (TC ≥ 50%) as determined by the VENTANA SP263 IHC assay, as assessed by central laboratories).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Must have at least 1 measurable lesion per RECIST v1.1
* Adequate organ and marrow function
* If a participant has brain or meningeal metastases, the participant must meet the following criteria:

  1. Have no evidence of progression by neurologic symptoms or signs for at least 4 weeks prior to the first dose.
  2. Participants with previously treated brain metastases may participate provided they have stable central nervous system (CNS) disease for at least 4 weeks prior to enrollment. Stable CNS disease is defined as resolution of all neurologic symptoms to baseline, having no evidence of new or enlarging brain metastases, and not requiring use of corticosteroids for CNS disease for at least 14 days prior to the start of study treatment. Participants who have had brain metastases resected or have received whole brain radiotherapy ending at least 4 weeks (or stereotactic radiotherapy ending at least 2 weeks) prior to initiation of study treatment are permitted.
  3. Carcinomatous meningitis is excluded regardless of clinical stability.

Key Exclusion Criteria:

* Presence of any tumor genomic aberration or driver mutation for which a targeted therapy is approved by local health authority and available
* Use of any live vaccines against infectious diseases within 28 days of first dose
* Any active autoimmune disease or a documented history of autoimmune disease or syndrome that required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs), except for vitiligo or resolved childhood asthma/atopy.
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or prostate cancer
* Prior treatment with any anti-PD-1, anti-PD-L1 or any other antibody targeting an immune checkpoint.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From randomization until death from any cause (up to 7 years)

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death from any cause (up to 7 years)
Confirmed Overall Response Rate (ORR) | From randomization until death from any cause (up to 7 years)
Number of Participants With treatment-emergent adverse events | From randomization until death from any cause (up to 7 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences, Inc.
Locations (92):
- Hope and Healing Cancer Service, Hinsdale, Illinois, United States
- Greece (4):
  - General hospital of Athens, chest diseases Sotiria, Athens
  - University General Hospital "Attikon", Chaïdári
  - General Oncology Hospital of Kifissia " Agioi Anargyroi", Kifissia
  - General Hospital of Patra Agios Andreas, Pátrai
- Hong Kong (5):
  - Hong Kong Integrated Oncology Centre, Hong Kong
  - Hong Kong United Oncology Centre, Hong Kong
  - Humanity and Health Clinical Trial Centre, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Malaysia (10):
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
  - Hospital Pulau Pinang, Pulau Pinang
  - Mount Miriam Cancer Hospital, Pulau Pinang
  - Institut Kanser Negara, Putrajaya
- Mexico (2):
  - Health Pharma Professional Research, Benito Juárez
  - Hospital Civil Fray Antonio Alcalde, Guadalajara
- Philippines (5):
  - Chong Hua Hospital, Cebu
  - Metro Davao Medical and Research Centre, Davao City
  - Makati Medical Centre, Manila
  - Philippine General Hospital, Manila
  - St. Luke Medical Centre Quezon City, Quezon City
- South Africa (7):
  - Exellentis Clinical Trial Consultants, George
  - Cancercare PE, Johannesburg
  - The Medical Oncology Centre of Rosebank, Johannesburg
  - Wits Clinical Research CMJAH Clinical Trial Site, Johannesburg
  - Port Elizabeth Oncology Centre-Cancercare, Port Elizabeth
  - University of Pretoria Medical Oncology, Pretoria
  - Wilgers Oncology Centre, Pretoria
- South Korea (18):
  - Dong-A University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - The Catholic University of Korea Incheon St. Mary's Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Cha University Bundang Medical Center, Seongnam
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital Yonsei University Health System, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Eunpyeong St. Mary's Hospital, Seoul
  - Ajou University Hospital., Suwon
  - The Catholic University of Korea St. Vincent Hospital, Suwon
  - Pusan National University Yangsan Hospital, Yangsan
- Taiwan (5):
  - Chang Gung Medical Foundation Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
- Thailand (19):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Police General Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Vajira Hospital, Bangkok
  - Saraburi Hospital, Changwat Sara Buri
  - Prapokklao Hospital, Chanthaburi
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Nakornping Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Lampang Hospital, Lampang
  - HRH Princess Maha Chakri Sirindhorn Medical Centre, Nakhon Nayok
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
  - Buddhachinaraj Phitsanulok Hospital, Phitsanulok
  - Naresuan University Hospital, Phitsanulok
  - Songkhlanagarind Hospital, Songkhla
  - Sunpasitthiprasing Hospital, Ubon Ratchathani
  - Udon Thani Hospital, Udon Thani
- Turkey (Türkiye) (13):
  - Adana City Hospital, Adana
  - Ankara City Hospital, Adana
  - Gazi University Medical Faculty, Ankara
  - Memorial Ankara Hospital, Ankara
  - Gazi University Medical Faculty, Çankaya
  - Trakya University Medical Faculty, Edirne
  - Acibadem Atakent Hospital, Istanbul
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Medipol University Medical Facility, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Kocaeli Universitiesi Tip Fakultesi, Kocaeli
  - Dicle University, Medical faculty, Sur
- Vietnam (3):
  - 103 Military Hospital, Hanoi
  - National Lung Hospital, Hanoi
  - Hue Central Hospital, Huế

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-10 - Public Website — https://trials.arcusbio.com/study/?id=ARC-10